## VAN YÜZÜNCÜ YIL UNIVERSITY DURSUN ODABAŞ MEDICAL CENTER INFORMED CONSENT FORM FOR RESEARCH

Dear patient,

Please read this document carefully and listen carefully to what we have said. Detailed information about the research; Detailed information about your rights, benefits and risks of the research can be found in this document. The purpose of these statements is to inform you about your health. Please indicate what you do not understand, your questions will be explained in detail. You can leave the research at any stage of the research if you think that your questions are not adequately explained after you accept to participate in the research or for any other reason. During the research period, the health problems arising from our research will be treated in our hospital immediately. You will not be charged an additional fee for participating in this research, nor will you be paid. Thank you for participating in our research.

Name of the Study: Comparison of I-Prf Impregnated Collagen with L-Prf in terms of Postoperative Complications and Wound Healing After Lower Impacted Third Molar Teeth Surgery

## The subject, purpose, method, time and process to be used of the research:

Our research is to examine the contribution of putting blood taken from the arm into the extraction socket of centrifuge products during the surgery of impacted wisdom teeth, to wound healing and patient comfort.

In the study, two types of plasma (I-PRF and L-PRF) will be obtained by centrifuging the blood taken from the arms of the patients. One of the plasmas (I-PRF) will be applied with type 1 collagen, and the other (L-PRF) alone will be applied to the extraction socket during the wisdom tooth operation at different times (there will be 5 weeks between both operations) Both surgical sites will be sutured with silk sutures

Check-ups will be made in the first session of the patients, on the 2nd and 7th days after the operation, and in the 2nd and 4th weeks. All patients after the operation; amoxicillin 500mg(Largopen 500mg, 3\*1), ibuprofen 600mg (Brufen 600 mg, 2\*1), benzydamine HcL + chlorhexidine gluconate mouthwash (Andorex 200ml mouthwash, 3\*1) will be used routinely. Sutures will be removed after 1 week. Postoperative complications will be evaluated in control sessions. Statistical analysis will be made and interpreted for the data obtained.

## Damages or possible risks that may occur during the research:

Risks of impacted tooth extraction and vascular access:

- 1. Swelling and/or redness, discomfort at the surgical site,
- 2. Redness and cracking in the corners of the mouth due to stretching,
- 3. Development of infection and delayed healing of the wound,
- 4. Dry socket; jaw pain that begins a few days after surgery, usually due to inadequate care; It is more common in lower jaw extractions, especially in wisdom teeth.
- 5. Damage to the adjacent tooth, breakage of the needle, especially in the presence of large fillings and crowns
- 6. Loss of sensation or decreased sensation in the gums, lips, tongue, teeth and jaw tip. It can be seen especially in teeth whose roots are close to the nerves, such as wisdom teeth. Numbness almost always returns to normal, but very rarely it can be permanent.
- 7. Trismus; It is a limitation in opening the mouth due to inflammation or swelling.
- 8. Bleeding-severe bleeding is not common. But bleeding in the form of leakage continues for several hours.
- 9. Sharp corners and bony steps may occur in the shooting cavities after extraction. These are corrected with a new surgical intervention.
- 10. Incomplete removal of root fragments. Sometimes small pieces of root can be left in order not to damage important formations such as sinuses or nerves.
- 11. Muscle relationship; The roots of the mandibular posterior teeth may be very close to the posterior tissue and muscle spaces, and in some cases, root fragments may escape into the cavity; These situations may require special attention or a second operation.

- 12. Jaw fractures; Although it is very rare, it is possible to occur in difficult and deeply impacted tooth extractions.
- 13. Extravasation of the needle, damage to the structures under the skin and around the vessel
- 14. Blood may collect around the needle site. (hematoma)
- 15. As a result of infection (germ catching), pain, redness, swelling may develop along the vein.
- 16. The development of a clot in the vein may cause the development of venous occlusion.
- 17. The needle may enter the artery and special effort may be required to stop the bleeding.
- 18. Air may enter the vein, resulting in an air plug. This plug can cause permanent disability.
- 19. Abscess, pain, bleeding, bruising, swelling and infection may develop in the area where the needle was inserted or in the operation area. Psychological process may develop. This situation may take time to improve.

Study-specific risks during the study: Allergic reaction

Signature:

Possible benefits of the research: The effectiveness of prf and i-prf-impregnated collagen plug on post-operative complications and wound healing will be determined after the impacted wisdom tooth surgery.

Anesthesia: Mandibular block anesthesia will be performed during the treatment.

Funding of the research: You will not be charged an additional fee for participating in this research

| and you will not be paid any money. | additional for for participating in this | 3 103041011 |
|---|---|---|
| Dear patient/ participant/fill in the relevant blank or tick the relevant box | ., please read the following articles car | efully and |
| 1. I was invited to the research after I received the prelimation a clear and simple way and after reading the consense I did not accept. | nt form in my hand. subject invitation; | I agreed. |
| 2. I have read and listened to the points to be considered research. Required enlightening answers don't understand. | ¥ <b>A</b> | about the I't get it, I |
| 3. Provided that my identity is kept confidential and us may be photographed during the intervention/treatmentercorectively or recorded. I allow I do not 4. I learned the benefits and possible risks of diagnostic | nt to be applied to me, that my data ca<br>allow. ———————————————————————————————————— | n be used reatments, |
| 6. The data received by me regarding the research will know. | be kept confidential, i know | i don't |
| 7. I have the right to withdraw from the research at any 8. I will not charge/pay any fee as a result of the research 9. If a medical risk arises, free medical treatment will be 10. The possible benefits of the research result in detail. 12. When I encounter a health problem during the remaind Mehmet GÜZEL at 05363609854 (mobile) and at YYU and Maxillofacial Surgery. | h; i know i don't know i don't know i don't know i know i don't know search; at any hour, Dt. I know that | ow I can call |
| The Participant's and/or Legal Representative to Get C | onsent in Emergency Situations | |
| Date: | Name-Surname of the Physic | ian |
| Phone. No: | Responsible for the Research | |
| Name surname: | Associate Professor Levent CİĞ | |
| Date of birth: | Institution Registration Number: 5086 | |
| Adress: | Signature: | |
| | ~ | |